CLINICAL TRIAL: NCT02024789
Title: A MULTI-CENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED PHASE 2 STUDY OF THE EFFICACY, SAFETY AND TOLERABILITY OF RG1662 IN ADULTS AND ADOLESCENTS WITH DOWN SYNDROME (CLEMATIS)
Brief Title: A Study of RG1662 in Adults and Adolescents With Down Syndrome (CLEMATIS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP27832; 2013-001263-23 (EudraCT Number)
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RG1662 120 mg bid (Experimental)
  Interventions: Drug: RG1662
- RG1662 240 mg bid (Experimental)
  Interventions: Drug: RG1662

INTERVENTIONS:
Drug: Placebo — Orally twice daily, 26 weeks
  Arms: Placebo
Drug: RG1662 — 120 mg (80 mg for subjects 12 and 13 years of age) orally twice daily, 26 weeks
  Arms: RG1662 120 mg bid
Drug: RG1662 — 240 mg (160 mg for subjects 12 and 13 years of age) orally twice daily, 26 weeks
  Arms: RG1662 240 mg bid

SUMMARY:
This multi-center, randomized, double-blind, 3-arm, parallel-group, placebo-controlled study will evaluate the efficacy and safety of RG1662 in adults and adolescents with Down syndrome. Subjects will be randomized to receive RG1662 either at low or high dose or placebo orally twice daily for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 12-30 years of age inclusive
* Clinical diagnosis of Down syndrome (trisomy 21) confirmed by chromosomal analysis (karyotyping)
* Males, or non-pregnant, non-lactating females. For females of childbearing potential, strict contraceptive prevention is required.
* Body-mass Index (BMI) 18-42 and 15-30 kg/m2 inclusive for adults and adolescents respectively
* Ability to complete the Clinical Evaluation of Language Fundamentals (CELF)-preschool 2 word classes task
* Subjects must have a parent, or other reliable caregiver who agrees to accompany the subject to all clinic visits, provide information about the subject as required by the protocol, and ensure compliance with the medication schedule
* Study participants must have sufficient language, vision and hearing to participate in study evaluations, as judged clinically by investigator

Exclusion Criteria:

* Subjects with a current DSM 5 diagnosis of any primary psychiatric diagnosis (including ASD or MDD)
* Subjects with a history of infantile spasms, of West syndrome, Lennox-Gastaut syndrome, Early Infantile Epileptic Encephalopathy or any treatment-refractory epilepsy associated with cognitive or developmental regression, of severe head trauma or CNS infections (e.g. meningitis)
* Subjects with a known or suspected clinical seizure event of any type within 24 months prior to screening
* Clinically relevant ECG abnormalities at screening or baseline; QTcF above 450 ms; personal or family history (first degree relatives) of congenital long QT syndrome
* Inadequate renal or hepatic function

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 173 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2016-05-04 (Actual); Study Completion 2016-05-04 (Actual)

PRIMARY OUTCOMES:
Cognition as assessed by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) sub-tests | 26 weeks
Adaptive behavior as assessed by the Vineland Adaptive Behavior Scales-II (VABS-II) standard scores | 26 weeks
Clinical global impression as assessed by Clinician Rated Global Improvement (CGI-I) scale | 26 weeks

SECONDARY OUTCOMES:
Incidence of abnormal ECG changes | 26 weeks
Abnormal ECG changes in adolescents as compared to baseline | from baseline to Week 26
Safety: Incidence of adverse events | approximately 32 weeks
Incidence of abnormal blood pressure | 26 weeks
RG1662 plasma concentrations | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- United States (9):
  - Univ of CA San Diego; Neurosciences Comp.Alzheimer's, La Jolla, California
  - University of California DAVIS Medical Center; M.I.N.D. Institute, Section of Developmental Behavior, Sacramento, California
  - Emory University School of Medicine; Department of Human Genetics & Pediatrics, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins Hospital., Baltimore, Maryland
  - Massachusette General Hospital; Medical Genetics, Boston, Massachusetts
  - Duke Clin Rsch Institute, Durham, North Carolina
  - University of Utah School of Medicine; Department of Pediatrics, Salt Lake City, Utah
  - University of Wisconsin Madison, Waisman Center, Madison, Wisconsin
- Argentina (2):
  - FLENI, CABA
  - Instituto Neurologia Bs As, Ciudad Autonoma de Bs As
- True North Clinical Research Kentville, Kentville, Nova Scotia, Canada
- France (4):
  - Groupement Hospitalier Est-Hopital Femme Mere enfant/Hospice civils de lyon, Bron
  - CHU de Montpellier Hopital Arnaud de Villeneuve; de Génétique, Montpellier
  - Institut Jérôme Lejeune; Neuropsychology, Paris
  - CHU de Saint Etienne; Service de Génétique, Saint-Etienne
- Italy (3):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Policlinico Universitario "Agostino Gemelli";Dip. Tutela Salute Donna Bambino Adolescente, Rome, Lazio
  - Ospedale Microcitemico; Clinica Pediatrica, Cagliari, Sardinia
- Mexico (4):
  - Hospital Dr. Angel Leaño; Pediatria, Guadalajara, Jalisco
  - Clínica Para la Atención del Neurodesarrollo, Aguascalientes
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez; Pediatria, Monterrey
  - Hospital Médica Tec 100, Querétaro
- New Zealand (3):
  - Auckland Clinical Studies, Auckland
  - University of Otago; Psychological Medicine Department, Dunedin
  - Wellington Hospital Research Office, Wellington
- KK Women's and Children's Hospital; Department of Neonatology, Singapore, Singapore
- Spain (6):
  - UVaMID Hospital Santa Caterina;; Servicio de Neurología, Salt, Girona
  - Complejo Hospitalario Universitario de Santiago (CHUS); Area Asistencial Integrada de Pediatría, Santiago de Compostela, La Coruña
  - IMIM, Human Pharmacology and Clinical Neurosciences,, Barcelona
  - Hospital Universitario de la Princesa; Medicina Interna, Madrid
  - Hospital Infantil Universitario Niño Jesus; Pediatria Social, Madrid
  - Fundación Síndrome de Down; Fundación Síndrome de Down, Madrid
- United Kingdom (4):
  - Blackpool Teaching Hospitals NHS Foundation Trust; Child Development and Family Support Centre, Blackpool
  - Mental Health of Learning Disability, Kent & Medway NHS and Social Care Partnership Trust, Dartford, Kent
  - Doncaster and Bassetlaw Hospitals NHS Foundation Trust; Doncaster Royal Infirmary, Doncaster
  - Cornwall Partnership NHS Foundation Trust, Redruth

REFERENCES:
- [Derived] Goeldner C, Kishnani PS, Skotko BG, Casero JL, Hipp JF, Derks M, Hernandez MC, Khwaja O, Lennon-Chrimes S, Noeldeke J, Pellicer S, Squassante L, Visootsak J, Wandel C, Fontoura P, d'Ardhuy XL; Clematis Study Group. A randomized, double-blind, placebo-controlled phase II trial to explore the effects of a GABAA-alpha5 NAM (basmisanil) on intellectual disability associated with Down syndrome. J Neurodev Disord. 2022 Feb 5;14(1):10. doi: 10.1186/s11689-022-09418-0. PMID 35123401